CLINICAL TRIAL: NCT07199959
Title: A Multi-center Retrospective Study of the Mechanism of Acquired Resistance in First Line Treatment of ROS1fusion Positive NSCLC With Entrectinib
Brief Title: Study on the Mechanism of Acquired Resistance of Entrectinib
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Ruijin Hospital (Other); The First Affiliated Hospital of Shanghai Jiaotong University (Unknown)
Responsible Party: Principal Investigator, Jialei Wang, Chief physician, Fudan University
Other Study IDs: EQTN-IIT-01
Record Dates: First submitted 2024-11-12; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: ROS1 Fusion Positive; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — entrectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood and tumor tissue
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: venipuncyure — venipuncture as clinical practical setting
Drug: Entrectinib — 600mg, oral, once daily

SUMMARY:
The goal of this observational study is to learn about the mechanism of acquired resistance in first line trearment of ROS1-positive NSCLC with entrectinib. The main question it aims to answer is:

what is the acquired resistant mechanism of entrectinib as first line treatment setting in patients?

Tissue or blood samples of participants who have already taken entrectinib as their regular medical care for NSCLC will send for Next gene sequencing for genomic profiles and bioinformatic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Histologically or cytologically diagnosed as non-small cell lung cancer (NSCLC);
* Clinically staged as IIIB-IV, unresectable locally advanced, recurrent, or metastatic NSCLC according to the 8th edition of the AJCC Lung Cancer Staging Manual;
* ROS1 fusion detected in tissue, cytological, or liquid biopsy specimens (such as plasma, cerebrospinal fluid, pleural effusion, or ascites) through molecular testing methods such as FISH, RT-PCR, NGS, etc.;
* At least one measurable lesion according to RECIST 1.1 criteria;
* No prior systemic anti-cancer treatment for locally advanced/metastatic disease (such as chemotherapy, targeted therapy, immunotherapy, anti-angiogenic therapy, etc.); patients who have previously received platinum-based adjuvant/neoadjuvant chemo/radiotherapy or radical chemo/radiotherapy for progressive disease are eligible if disease progression occurs more than 6 months after the last treatment;
* For patients who have progressed on first-line treatment with entrectinib and have tissue specimens or peripheral blood samples before and after treatment with entrectinib, they may participate in this study;
* For patients who are currently on first-line treatment with entrectinib and have not yet progressed, if they have tissue specimens or peripheral blood samples before treatment with entrectinib and agree to participate in this study and sign an informed consent form to collect tissue specimens or peripheral blood samples at the time of first treatment follow-up progression, they may participate in this study;
* For newly diagnosed patients who have not yet received any drug treatment, those who need first-line treatment with entrectinib according to the clinical standard of care, after agreeing to participate in this study and signing an informed consent form, will have tissue specimens or peripheral blood samples collected before treatment with entrectinib, followed by routine drug use and treatment follow-up, and additional tissue specimens or peripheral blood samples will be collected at the time of first treatment follow-up progression;
* Cooperate with the researchers to provide clinical and pathological data, imaging data, biological specimen collection, follow-up, etc., required for the study process, and agree to use the testing data for this study.

Exclusion Criteria:

* Patients with mixed small cell lung cancer components.
* Carrying other clearly druggable targets, such as EGFR sensitive mutations, EGFR exon 20 insertions, ALK fusions, RET fusions, KRAS activating mutations, BRAF V600E mutations, NTRK1/2/3 fusions, ERBB2 exon 20 insertions, MET exon 14 skipping, MET amplification, etc.
* Having received prior systemic treatment (such as chemotherapy, targeted therapy, immunotherapy, anti-angiogenic therapy, etc.).
* Suffering from other malignant tumors within the past 5 years, with the exception of those with very low risks of metastasis or death (5-year RFS rate > 90%, such as early-stage prostate cancer, breast cancer, etc.).
* Having any contraindications to entrectinib treatment.
* Being unable to understand the informed consent form, unable to cooperate with sample collection and follow-up, or refusing to sign the informed consent form.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinically staged as IIIB-IV, unresectable locally advanced, recurrent, or metastatic ROS1 fusion positive non small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
biomarker profile | Analysis will occur when all patient samples have collected. From enrollment to the study completion, an average of 2 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university shanghai cancer center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided